CLINICAL TRIAL: NCT02007239
Title: Cytokine Blockade With Tocilizumab in Patients With Cytokine Release Syndrome and Hemophagocytic Lymphohistiocytosis
Brief Title: Tocilizumab and Hemophagocytic Lymphohistiocytosis (HLH)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No subjects were enrolled
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-010459
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Hemophagocytic Lymphohistiocytosis
Keywords: tocilizumab; hemophagocytic lymphohistiocytosis (HLH); cytokine; cytokine release syndrome
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Cytokine Release Syndrome | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): single dose of tocilizumab (8mg/kg intravenously) within 24 hours of administration of standard immunochemotherapy.
  Interventions: Drug: tocilizumab

INTERVENTIONS:
Drug: tocilizumab — single dose of tocilizumab (8mg/kg intravenously) within 24 hours of administration of standard immunochemotherapy.
  Other Names: TCZ

SUMMARY:
This study seeks to determine the efficacy of tocilizumab (TCZ) in patients with hemophagocytic lymphohistiocytosis (HLH) and high cytokine levels (proteins involved in inflammation) in an attempt to decrease the damage caused by these proteins; and secondarily to assess its safety and impact on disease activity.

DETAILED DESCRIPTION:
Subjects with hemophagocytic lymphohistiocytosis (HLH) often have life-threatening complications at the time of diagnosis resulting from excessive inflammation. This excessive inflammation is driven by abnormally high levels of cytokines--proteins involved in inflammation. Standard therapy for HLH does not directly target these cytokines. Tocilizumab is a medicine that blocks one of the cytokines that is elevated in patients with HLH.

This is an open-label single-arm uncontrolled trial with biologic endpoint. This study will use tocilizumab in subjects with HLH and high cytokine levels in an attempt to decrease the damage caused by these proteins. All subjects will receive standard therapy, in addition to tocilizumab. We hypothesize the tocilizumab will decrease levels of certain important cytokines. This may make it easier to treat subjects with HLH overall.

TCZ will be administered as a single dose (8mg/kg) intravenously. Eligible subjects will be inpatients at the Children's Hospital of Philadelphia (CHOP) main campus. 10 subjects with HLH will be enrolled. All subjects will be initiated on standard HLH-directed treatment. Cytokine levels [including serum interferon (IFN-γ) and interleukin (IL-6)] will be monitored, in addition to other laboratory and clinical markers of HLH disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 3 months to 25 years.
2. Fulfill the clinical diagnostic criteria for HLH, as defined by the Histiocyte Society (see Table 1). Only patients with de novo HLH are eligible.
3. Evidence of cytokine release syndrome (CRS), as defined by EITHER:

   i. Known elevated interferon-γ and interleukin-6 ≥2x ULN, OR ii. If cytokine levels are unknown at the time of study enrollment:

   a. Fever of at least 38.5º celsius at minimum of once every 24 hours for at least 48 hours, AND either i. Respiratory insufficiency requiring oxygen supplementation of at least 2 Liter by nasal cannula for at least 12 hours (also including invasive, noninvasive, continuous positive airway pressure or biphasic airway pressure for the purpose of treating respiratory failure), OR ii. Vasoactive infusion for at least 12 hours, including dopamine ≥5mcg/kg/min, dobutamine≥5mcg/kg/min, or any dose of epinephrine, norepinephrine, milrinone, or vasopressin.
4. Patients must be planned to initiate HLH-directed therapy within 24 hours of study enrollment.
5. Girls >= 11 years of age must have a negative urine/serum pregnancy test and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
6. Parental/guardian permission (informed consent)

Exclusion Criteria:

1. On-going or planned participation in another clinical trial involving HLH-directed treatment
2. Previous administration of any other biologic agent targeted at cytokine blockade within 5 days of enrollment.
3. Renal insufficiency defined by estimated glomerular filtration rate (based on modified Schwartz formula) <50 ml/min, or need for renal replacement therapy.
4. Hepatic dysfunction as defined by serum alanine aminotransferase (ALT)>=10x upper limit of normal (ULN). For the purposes of this study, the ULN for ALT is 45 U/L.
5. HLH that is relapsed, refractory, or considered to be therapy-related, as in the case of T cell-activating therapies.
6. Established prior diagnosis of underlying rheumatologic condition, including juvenile idiopathic arthritis.
7. Pregnant or lactating females.
8. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
9. Suspected gastrointestinal perforation.
10. Known or suspected demyelinating central nervous system disease.
11. Known history of tuberculosis.
12. Transfusion-refractory thrombocytopenia defined as inability to maintain platelet count over 30,000/ul for at least 6 hours with transfusion support.
13. Known active herpetic infection.
14. Inability to start HLH-directed immunochemotherapy.

Ages: 3 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Reduction in serum interferon-gamma levels after tocilizumab (TCZ) administration | baseline, 24 -36 hours, and 4-7 days after administration of TCZ
  Assess change in interferon gamma levels from the screening visit to the measurements taken within 24-36 hours and at 4-7 days after drug administration.

SECONDARY OUTCOMES:
Change in other cytokine levels (interleukin-6, interleukin-10, tumor necrosis factor-alpha, etc.) | baseline, 24-36 hour, then weekly for 4 weeks after administration of TCZ
  Cytokine levels [IL-1, IL-2, sIL-2r, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, IL-13, Tumor necrosis factor-alpha (TNF-α) and IFN-γ] will be assessed at baseline, within 24-36 hours, then weekly for 4 weeks after TCZ administration;
Presence of HLH disease activity for each subject following TCZ administration | within 1 week of administration of TCZ
  HLH disease activity markers will be assessed for each subject (fever, ferritin, cardiopulmonary support requirements, cytopenias, coagulation tests, etc.)
Degree of hepatic function, cytopenias and infection in subjects following administration of TCZ | up to 1 year of administration of TCZ
  Degree of hepatic function, presence (or absence) of cytopenia/infection will be assessed based on changes in laboratory and clinical markers following administration of TCZ.
Overall survival of subjects | day 100 and survival to completion of therapy (blood/marrow transplant, if applicable)
  Overall survival of subjects will include survival to day 100, and survival to completion of therapy (HSCT for primary HLH, and end of induction therapy for secondary HLH).

CONTACTS AND LOCATIONS:
Overall Officials: David Teachey, MD, Principal Investigator — Division of Oncology, Department of Pediatrics, Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Henter JI, Samuelsson-Horne A, Arico M, Egeler RM, Elinder G, Filipovich AH, Gadner H, Imashuku S, Komp D, Ladisch S, Webb D, Janka G; Histocyte Society. Treatment of hemophagocytic lymphohistiocytosis with HLH-94 immunochemotherapy and bone marrow transplantation. Blood. 2002 Oct 1;100(7):2367-73. doi: 10.1182/blood-2002-01-0172. PMID 12239144
- [Background] Tang Y, Xu X, Song H, Yang S, Shi S, Wei J, Pan B, Zhao F, Liao C, Luo C. Early diagnostic and prognostic significance of a specific Th1/Th2 cytokine pattern in children with haemophagocytic syndrome. Br J Haematol. 2008 Oct;143(1):84-91. doi: 10.1111/j.1365-2141.2008.07298.x. Epub 2008 Jul 31. PMID 18673367
- [Background] Navarro-Millan I, Singh JA, Curtis JR. Systematic review of tocilizumab for rheumatoid arthritis: a new biologic agent targeting the interleukin-6 receptor. Clin Ther. 2012 Apr;34(4):788-802.e3. doi: 10.1016/j.clinthera.2012.02.014. Epub 2012 Mar 22. PMID 22444783
- [Background] Teachey DT, Rheingold SR, Maude SL, Zugmaier G, Barrett DM, Seif AE, Nichols KE, Suppa EK, Kalos M, Berg RA, Fitzgerald JC, Aplenc R, Gore L, Grupp SA. Cytokine release syndrome after blinatumomab treatment related to abnormal macrophage activation and ameliorated with cytokine-directed therapy. Blood. 2013 Jun 27;121(26):5154-7. doi: 10.1182/blood-2013-02-485623. Epub 2013 May 15. PMID 23678006
- [Background] Grupp SA, Kalos M, Barrett D, Aplenc R, Porter DL, Rheingold SR, Teachey DT, Chew A, Hauck B, Wright JF, Milone MC, Levine BL, June CH. Chimeric antigen receptor-modified T cells for acute lymphoid leukemia. N Engl J Med. 2013 Apr 18;368(16):1509-1518. doi: 10.1056/NEJMoa1215134. Epub 2013 Mar 25. PMID 23527958